CLINICAL TRIAL: NCT07155863
Title: The Effect of Ear Plugs and Eye Patch on Anxiety Level During Magnetic Resonance Imaging
Brief Title: The Effect of Sensory Isolation on Anxiety in Magnetic Resonance Imaging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Saadet Saza, Specialist Nurse, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ege-SBF-SS-01
Record Dates: First submitted 2025-08-14; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Thorax Injuries; Cervical Injury Spine; Brain Trauma; Joint Trauma
Keywords: Manyeyic resonance imagining; anxiety; noise; earplug; eye mask
MeSH Terms: conditions — Thoracic Injuries; Brain Injuries, Traumatic; Anxiety Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel- group study with 2 arms: an intervention group receiving earplugs and eye mask during MRI, and a control group receiving standard care without sensory isolation devices.
Who Masked: Outcomes Assessor
Masking Description: A single-blind method will be used to reduce bias in the study. The evaluator, who will record physiological indicators (pulse, blood pressure, saturation value) and apply the anxiety scale, will not know which group the participants belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Earplugs ve eye mask Arm (Experimental): The patient information form containing the patient's pre-imaging information, anxiety monitoring form, and physiological symptoms will be measured and recorded as necessary. The researcher will provide a brief explanation about the imaging procedure to the intervention group, and each individual will be given a single-use earplug and eye mask to wear during the imaging procedure. Immediately after the imaging procedure, the anxiety monitoring form will be completed again, and physiological symptoms will be measured and recorded.
  Interventions: Device: Earplugs and eye mask
- 2. Control Arm (No Intervention): Participants in the control group will receive standard care without any additional experimental intervention. Physiological parameters and anxiety levels will be assessed at baseline and the end of the imaging.

INTERVENTIONS:
Device: Earplugs and eye mask — Participants in the experimental group will use earplugs and eye mask during MRI. The use of these devices aims to decrease anxiety levels caused by noise and the MRI procedure. Physiological parameters and axiety scores will be monitored throughout the study.
  Arms: 1. Earplugs ve eye mask Arm

SUMMARY:
The aim of this study is to determine whether the use of earplugs and eye masks in adults reduces anxiety during Manyetic Resonance Imaging. In addition, in order to evaluate the effect of earplugs and eye masks on the physiological symptoms of anxiety, the pulse rate, blood pressure, respiratory rate, and saturation value of adults will be measured before and after imaging.

H0: Earplugs and eye masks have no effect on state anxiety levels. H1: Earplugs and eye masks have an effect on state anxiety levels. H2: Earplugs and eye masks have an effect on heart rate. H3: Earplugs and eye masks have an effect on respiratory rate. H4: Earplugs and eye masks have an effect on systolic blood pressure. H5: Earplugs and eye masks have an effect on diastolic blood pressure. H6: Earplugs and eye masks have an effect on saturation values.

DETAILED DESCRIPTION:
Patients who have previously had appointments at the MR unit of Manisa Celal Bayar University Hafsa Sultan Hospital will be included in the study. In addition to the routine information provided by the MR technician to patients in the study group selected by random sampling, written consent (Informed Consent Form) will be obtained from patients who agree to participate in the study prior to MRG. The patient information form, anxiety monitoring form, and measurements of blood pressure, pulse rate, respiratory rate, and saturation rate will be recorded in the physiological signs section. Prior to imaging, the researcher will provide a brief explanation of the imaging process, and the participant will be provided with customised earplugs and an eye mask to wear during imaging. After imaging, blood pressure, pulse rate, respiratory rate, and saturation values will be measured again at 0 minutes, and the anxiety monitoring form will be completed. For the control group, written consent (Informed Consent Form) will be obtained from participants who have agreed to voluntarily participate in the study. Blood pressure, heart rate, respiratory rate, and oxygen saturation will be measured before and after the imaging, and no intervention will be performed. The study will include patients aged 18-65 who are participating in MRI for the first time, who have voluntarily agreed to participate in the study, and who have undergone brain, thoracic, and cervical MRI scans lasting at least 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Those who are undergoing an MRI scan for the first time,
* Those undergoing a scheduled MRI scan (emergencies will not be accepted)
* Those who are willing to participate in the study,
* MRI scans lasting at least 30 minutes,
* Those who are able to communicate verbally,
* Those who are not hospitalised are eligible for inclusion.

Exclusion Criteria:

* Those under 18 and over 65 years of age
* Patients who cannot tolerate MRI scans (those who require sedation/medication during the scan
* Patients with hearing or vision impairments,
* Pregnant or breastfeeding individuals,
* Individuals with severe comorbidities,
* Individuals with acute/chronic pain who are using analgesics,
* Individuals who cannot wear earplugs or eye patches (e.g., those with active ear infections, eye infections, or phobias),
* Individuals who refuse to participate in the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
''Change in Systolic Blood Pressure Before and After Magnetic Resonance Imaging'' | Pre- intervention and immediately after the intervention. ''Before MRI and immediately after MRI''
  Systolic blood pressure measured in seated position using an automated cuff. Change calculated as post-MRI minus pre-MRI.
  Measure Type/ Unit: mmHg
''Change in Diastolic Blood Pressure Before and After MRI'' | ''Before and immediately after MRI''
  Diastolic blood pressure measured in seated position with an automated cuff. Change is calculated as post MRI minus pre-MRI.
  Measure Type/unit: mmHg

SECONDARY OUTCOMES:
''Change in Heart Rate Before and after MRI'' | ''Post-MRI minus pre-MRI'' Measure Type/unit: bpm
  Heart rate measured via pulse oximetry; change is post MRI minus pre-MRI
''Change in Oxygen Saturation (SpO₂) Before and After MRI'' | ''Before MRI and immediately after MRI''
  Oxygen saturation is measured with a pulse oximeter and the unit is bpm.
''Change in State- Anxiety Inventory (STAI-I)'' | Pre- intervention and immediately after the intervention ''before MRI and immediately after MRI''
  The State Anxiety Inventory is a measurement tool consisting of statements that describe how a person feels at a particular moment, while the Trait Anxiety Inventory is a measurement tool consisting of statements that describe how a person generally feels.The State-Trait Anxiety Inventory is a self-assessment inventory consisting of short statements. Items 3, 4, 6, 7, 9, 12, 13, 14, 17, 18 items are assigned positive scores (increasing the total anxiety score), while items 1, 2, 5, 8, 10, 11, 15, 16, 19, 20 are assigned negative scores (decreasing the total anxiety score). When evaluating, a score between 1 (or -1) and 4 (or -4) is given for each item according to its positive or negative characteristic, and a constant of 50 should be added to the total score obtained. The highest possible score is 80, and the lowest is 20.
  Measure Type/Unit: point.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cevik K, Cetinkaya A, Yigit Gokbel K, Menekse B, Saza S, Tikiz C. The Effect of Abdominal Massage on Constipation in the Elderly Residing in Rest Homes. Gastroenterol Nurs. 2018 Sep/Oct;41(5):396-402. doi: 10.1097/SGA.0000000000000343. PMID 30272602
- See also: Related Info — https://bmcpsychiatry.biomedcentral.com/articles/10.1186/s12888-024-06091-6#citeas
- Available data/document: Study Protocol — https://bmcpsychiatry.biomedcentral.com/articles/10.1186/s12888-024-06091-6